CLINICAL TRIAL: NCT00134342
Title: A Comparison of Traditional Tuberculosis Screening Methods With the T-SPOT TB Test for the Diagnosis of Latent Tuberculosis Infection in Immunocompromised Populations
Brief Title: Tuberculosis (TB) Screening for the Diagnosis of Latent TB in Immunocompromised Populations
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Oxford Immunotec (Industry)
Responsible Party: Nial Ferguson, Oxford Immunotec
Other Study IDs: 04-0702-AE
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2010-12-23 (Estimated); Status verified 2005-07

CONDITIONS: Tuberculosis
Keywords: tuberculosis; tuberculin test; immunologic tests; Latent tuberculosis; end stage renal disease; solid organ transplantation; bone marrow transplantation; rheumatologic disease
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis; Kidney Failure, Chronic; Collagen Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: T-SPOT TB ELISPOT test — ELISPOT test for detecting T cell responses to tuberculosis antigens.

SUMMARY:
The tuberculin skin test (TST) has been the gold standard for diagnosing latent tuberculosis for almost 100 years. While this test performs reasonably well in healthy, non-bacille Calmette-Guerin (BCG) vaccinated populations, it is believed to perform less well in patients who do not have intact cellular immune systems (immunocompromised).

The investigators hypothesize that a new test, the T-SPOT TB ELISPOT test will provide a more accurate measurement of latent infection in immunocompromised people. This study will compare the TST to the T-SPOT TB ELISPOT test, and to the results of an expert physician diagnostic panel.

DETAILED DESCRIPTION:
Main Study Question:

We propose to investigate the correlation between the traditional TST-based method of screening for latent tuberculosis infection in specific immunocompromised populations as recommended by Canadian and American standards: the T-SPOT TB ELISPOT test: and an expert tuberculosis physician panel incorporating the Mantoux test, a risk factor survey, and a chest radiograph.

Secondary Study Question:

In a subset of patients who have tested positive on both the Mantoux and T-SPOT ELISPOT tests prior to undergoing additional immune suppression i.e., patients pre-bone marrow transplant and rheumatology patients pre-receipt of anti-TNF alpha therapy or high dose corticosteroids, we propose to repeat the T-SPOT ELISPOT and Mantoux after immune suppression to assess the development of cutaneous anergy.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the study are broad.

* Participants can be enrolled regardless of race, gender, risk of exposure to TB, metabolic disorders or coinfection with non-TB agents.
* Only participants who have provided written informed consent will be included.
* Patients belonging to the four following groups will be considered eligible for tuberculosis screening and inclusion in the T-SPOT ELISPOT study:

  * Patients with end stage renal disease receiving hemodialysis or peritoneal dialysis;
  * Recipients of solid organ transplants;
  * Recipients of, or candidates for, an allogeneic stem cell transplant for hematologic malignancies;
  * Patients with rheumatologic diseases (e.g., systemic lupus erythematosus [SLE], rheumatoid arthritis, psoriasis) who are receiving, or about to receive, immunosuppressive therapy, including corticosteroids and anti-TNF alpha inhibitors.

Exclusion Criteria:

* Individuals who have not signed an informed consent
* Hemophiliacs or individuals who, on the advice of the enrolling physician, may otherwise be at increased risk of an adverse reaction to venipuncture or tuberculin skin test administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with endstage renal disease
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2005-01; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gardam, MD, Principal Investigator — University Health Network, University of Toronto
Locations (2):
- Canada (2):
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario